CLINICAL TRIAL: NCT01850511
Title: The Effect of Vibrissae on Subjective and Objective Measures of Nasal Obstruction
Brief Title: The Effect of Nasal Hair on Nasal Obstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Grant S. Hamilton, III, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-001362
Record Dates: First submitted 2013-05-03; First posted 2013-05-09 (Estimated); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Nasal Obstruction
Keywords: Nasal obstruction; Vibrissae; Nasal hair
MeSH Terms: conditions — Nasal Obstruction | interventions — Oxymetazoline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vibrissae trimming (Experimental): Patients will serve as their own control, with assessment of primary outcomes pre- and post-trimming of vibrissae.
  Interventions: Procedure: Vibrissae trimming; Drug: Application of oxymetazoline

INTERVENTIONS:
Procedure: Vibrissae trimming — Patients will have oxymetazoline administered prior to assessment of outcome measures to ensure minimal impact of erectile mucosal tissue on measurement.
Drug: Application of oxymetazoline — Afrin will be administered to minimize the impact of erectile mucosal tissue on obstruction.
  Other Names: Afrin

SUMMARY:
Nasal obstruction is a common complaint prompting presentation to an otolaryngologist. Many studies have been performed quantifying and describing the impact of a number of factors on symptoms of nasal obstruction, including anatomical, neoplastic, infectious, and inflammatory causes. Despite this scrutiny, no attention has been paid to the nasal vibrissae as a potential anatomical contributor to nasal obstruction. The proposed study intends to elucidate that contribution, if any exists.

ELIGIBILITY:
Inclusion Criteria:

* Presence of nasal vibrissae
* Able to tolerate rhinomanometry

Exclusion Criteria:

* Anatomical or other obvious cause of obstruction
* Claustrophobia with rhinomanometry mask

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-05; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Nasal airflow/pressure | Participants will undergo assessment over a 30 minute period, no follow-up
  Objective measures include airflow and pressure as assessed by Rhinomanometry.
Subjective Nasal Obstruction | Participants will undergo assessment over a 30 minute period, no follow-up
  Subjective measures will be assessed via the modified version of the NOSE outcome instrument-a validated test of subjective nasal obstruction

CONTACTS AND LOCATIONS:
Overall Officials: Grant Hamilton, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Background] Ozturk AB, Damadoglu E, Karakaya G, Kalyoncu AF. Does nasal hair (vibrissae) density affect the risk of developing asthma in patients with seasonal rhinitis? Int Arch Allergy Immunol. 2011;156(1):75-80. doi: 10.1159/000321912. Epub 2011 Mar 30. PMID 21447962
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials